CLINICAL TRIAL: NCT04267250
Title: A PHASE 1, RANDOMIZED, OPEN LABEL, 2-WAY CROSSOVER STUDY TO ESTIMATE THE EFFECT OF MULTIPLE DOSE PF-06700841 ON THE PHARMACOKINETICS OF SINGLE DOSE ORAL CONTRACEPTIVE STEROIDS IN HEALTHY FEMALE PARTICIPANTS
Brief Title: Effect Of Multiple Dose PF-06700841 On The Pharmacokinetics Of Single Dose Oral Contraceptive Steroids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7931018; Oral Contraceptive DDI (Other: Alias Study Number)
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Healthy Female Volunteers
MeSH Terms: interventions — PF-06700841; Ethinyl Estradiol; Levonorgestrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): In sequence 1, period 1, participants will be dosed with a single administration of oral contraceptive (OC). Participants will continue directly into period 2 where they will receive PF-06700841 PO for 13 days with a single dose of OC administered on the morning of day 10.
  Interventions: Drug: PF-06700841; Drug: Ethinyl estradiol (EE) and levonorgestrel (LN)
- Sequence 2 (Experimental): In sequence 2, period 1, participants will receive PF-06700841 PO for 13 days with a single dose of OC administered on the morning of day 10. After a wash-out period of at least 10 days, participants will continue into period 2 where they will receive an additional single dose of OC.
  Interventions: Drug: PF-06700841; Drug: Ethinyl estradiol (EE) and levonorgestrel (LN)

INTERVENTIONS:
Drug: PF-06700841 — 60 mg by mouth (PO) once daily (QD).
Drug: Ethinyl estradiol (EE) and levonorgestrel (LN) — Oral tablet containing 30 mcg EE and 150 mcg LN.

SUMMARY:
This Phase 1 study will assess the pharmacokinetic effect of multiple doses PF 06700841 (administered once a day) on a single dose of a combination oral contraceptive, in 18 healthy female participants who are not of childbearing potential.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, 2 way crossover, multiple-dose, open label study of the effect of multiple doses PF-06700841 on single dose combination oral contraceptive (OC) pharmacokinetics (PK) in healthy female participants aged 18-60.

The study consists of a screening phase (up to 28 days prior to Day 1); two treatment periods during which participants are resident in the Clinical Research Unit (CRU) and a final follow-up telephone contact, which will be conducted after 28-35 following administration of the last dose.

Participants will be randomized to 1 of 2 treatment sequences. A total of 18 healthy female participants (9 in each treatment sequence) will be enrolled in the study. Each treatment sequence will consist of 2 periods in a single fixed sequence. Participants will be screened within 28 days of the first dose of investigational product. Participants will report to the Clinical Research Unit (CRU) the day prior to Day 1 dosing in Period 1 for both treatment sequences, and will report to the CRU the day prior to Day 1 dosing in Period 2 for Treatment Sequence 2. In Treatment Sequence 1, participants will remain in the CRU for up to 21 days and 20 nights. There will be no washout period in Treatment Sequence 1. In Treatment Sequence 2, participants will remain in the CRU for up to 22 days and 20 nights. Participants in treatment sequence 2 will have an outpatient washout period of at least 10 days between Period 1 and Period 2. A single administration of OC in the form of 1 PORTIA or equivalent tablet will be administered in one of the two periods (reference treatment) and in the alternative treatment period, daily doses of 60 mg PF-06700841 will be administered for 13 days with a single dose of OC being administered on Day 10. PK (AUCinf, Cmax, AUClast, Tmax and t½) of OC will then be assessed at pre OC dose and over 96 hours, post OC dosing.

Safety assessments will be conducted at the CRU.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females aged 18-60
* Not of childbearing potential
* Body mass index of 17.5-30.5 kg/m2
* Body weight > 50 kg
* Capable of giving signed informed consent

Exclusion Criteria:

* Evidence or history of clinically significant disease including irritable bowel disease; HIV; Hep B and Hep C; acute or chronic infection history; lymphoproliferative disorder; tuberculosis; hearing loss; sensitivity to heparin or heparin-induced thrombocytopenia
* Any condition affecting drug absorption
* Participants who have experienced major trauma or surgery in the 3 months prior to baseline
* Participants in imminent need for surgery
* Use of prescription or non-prescription drugs within 7 days or 5 half-lives prior to dosing
* Previous administration with an investigational drug within 30 days or 5 half-lives prior to dosing
* A positive urine drug test
* Hypertension
* ECG anomalies
* Significant laboratory anomalies
* History of drug abuse with less than 6 months of abstinence prior to the baseline visit
* History of alcohol abuse within 6 months of screening
* History of nicotine use within 30 days of baseline visit
* Any contraindications to OC
* History of discontinued use of OC for medical reasons
* Febrile illness within 5 days prior to dosing
* Vaccination with live or attenuated virus or live viral components within 6 weeks prior to dosing
* History of major organ transplant
* History of severe allergic or anaphylactic reaction to kinase inhibitors
* have donated blood of 500mL or more within 60 days prior to dosing

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for EE | 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post OC dose in periods 1 and 2
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for LN | 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post OC dose in periods 1 and 2
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Quotient Sciences Screening Office, Coral Gables, Florida
  - Quotient Sciences-Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7931018